CLINICAL TRIAL: NCT00666055
Title: CID 0708 - Sex, Aging and Antiretroviral Pharmacokinetics
Brief Title: Sex, Aging and Antiretroviral Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: Kristine Patterson, MD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Kristine Patterson, MD, Clinical Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: CID 0708; 1K23AI077355-01 (NIH)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Sex; Aging; Antiretroviral; Pharmacokinetics; post-menopausal women with HIV infection; pre-menopausal women with HIV infection
MeSH Terms: conditions — HIV Infections; Coitus | interventions — Zidovudine; Lamivudine; Emtricitabine; Tenofovir; efavirenz; Lopinavir; lopinavir-ritonavir drug combination; Atazanavir Sulfate; Ritonavir; Maraviroc; Raltegravir Potassium; etravirine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood; genital secretions; genital tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 30 post-menopausal HIV-infected women
  Interventions: Drug: ARV regimen chosen by treating physician
- Group 2: 12 pre-menopausal HIV-infected women
  Interventions: Drug: ARV regimen chosen by treating physician

INTERVENTIONS:
Drug: ARV regimen chosen by treating physician — Women may also be naïve to either NNRTI or PIs and initiating their first, second or third HAART regimen (ARVs to be investigated: zidovudine, lamivudine, emtricitabine, abacavir, tenofovir, efavirenz, lopinavir/ritonavir, atazanavir with or without ritonavir).
  Provided the ARV regimens contain one or more of the agents under study they may also include new agents such as maraviroc (CCR5 inhibitor), raltegravir (integrase inhibitor) and/or etravirine (NNRTI).
  Other Names: Zidovudine: ZDV, Retrovir, Retrovis, AZT (Azidothymidine); Lamivudine: 3TC, Zeffix, Epivir, Epivir-HBV; Emtricitabine: FTC, Emtriva; Abacivir: Ziagen; Tenofovir: TDF, Viread; Efavirenz: Sustiva, Stocrin; Lopinavir/Ritonavir: Kaletra, Aluvia; Atazanavir: Reyataz; Ritonavir: Norvir; Maraviroc: Selzentry; Raltegravir: MK-0518, Isentress; Etravirine: TMC-125, Intelence

SUMMARY:
The purpose of this research study is to learn about levels of antiretroviral drug levels and response to HIV virus in the genital tract of women who are post-menopausal. The investigators in this study think that the levels of hormones post-menopausal HIV-infected women may have in their bodies may affect the levels of antiretroviral drug, and therefore affect how much HIV virus they have in their bodies. Since women who have already gone through menopause have different levels of hormones, such as estrogen, than women who are pre-menopausal, the investigators would like to check the levels of antiretroviral drugs in their blood, their genital secretions, and their genital tissue.

DETAILED DESCRIPTION:
Purpose: To longitudinally quantify systemic and genital tract antiretroviral pharmacokinetics and viral responses in HIV-infected post-menopausal women. These parameters will be compared to pre-menopausal women to determine if the absence or presence of estrogen influences treatment responses and infectiousness of HIV.

Participants: 30 post-menopausal and 12 pre-menopausal HIV-infected women Procedures (methods): First dose, steady state, and longitudinal pharmacokinetics of the most commonly prescribed antiretroviral agents will be assessed in the systemic and genital tract compartments in a cohort of post- and pre-menopausal HIV-infected women. Concurrent blood plasma and genital secretions HIV RNA will be measured. Systemic and genital tract virologic responses will be correlated with antiretroviral concentrations and with each other.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected women >18 years of age
2. There are no specific entry criteria for CD4+ T-cell counts and plasma HIV RNA.
3. Menopause status will be determined at screening.

   1. Post-menopausal will be defined as the cessation of menses for >12 months (or undergone a bilateral oophorectomy with or without a hysterectomy) AND a FSH >25 miu/mL and estradiol level <20 pg/mL establishing both physiological and biochemical evidence of menopause.
   2. Pre-menopausal women must have regular cycles without peri-menopausal vasomotor symptoms and not receiving exogenous hormones.
4. Women may be changing to a new regimen because of virologic failure or intolerability. Women in whom resistance testing is available, two or more drugs to which the virus is susceptible needs to be included in the proposed treatment regimen.
5. Women may also be naïve to either NNRTI or PIs and initiating their first, second or third HAART regimen (ARVs to be investigated: zidovudine, lamivudine, emtricitabine, abacavir, tenofovir, efavirenz, lopinavir/ritonavir, atazanavir with or without ritonavir).
6. Provided the ARV regimens contain one or more of the agents under study they may also include new agents such as maraviroc (CCR5 inhibitor), raltegravir (integrase inhibitor) and/or etravirine (NNRTI). Samples will be stored so that the pharmacokinetics of these agents can be evaluated in future studies once the assays are available in our lab.
7. Women must be free from sexually transmitted infections (STI's) at the time of enrollment.
8. Women must be able to abstain from douching and sexual activity for 72 hours prior to all study visits.
9. Subjects must be willing to have genital tract samples taken.

Exclusion Criteria:

1. Women currently receiving medication with known drug-drug interaction with the ARVs under study.
2. Women currently receiving any exogenous hormone therapy (contraception, estrogen replacement therapy or androgen supplements). Women must be off all exogenous hormone therapy for > 16 weeks prior to enrollment.
3. Women who are pregnant or breast-feeding.
4. Women with a hemoglobin <9.0g/dL and/or hematocrit <28%.
5. Women unable to complete, or have a caretaker complete, a dose administration card.
6. Women who, in the judgement of the investigator, are unable to comply with the protocol requirements.
7. Women who are unable to give written informed consent.
8. Women who cannot comply with abstaining from intercourse or douching 48 hours prior to study examination.
9. Male or transgender individuals.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will primarily be recruited from the UNC Infectious Disease Clinic and the Wake County HIV Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To measure and compare steady state blood plasma pharmacokinetics of antiretroviral therapies in post- and pre-menopausal HIV-infected women. | 6 months

SECONDARY OUTCOMES:
To longitudinally quantify and compare genital tract antiretroviral drug exposure in post- and pre-menopausal HIV-infected women | 6 months
To determine and compare sexual HIV infectivity in post- and pre-menopausal HIV-infected women by measuring HIV RNA dynamics in blood plasma and genital tract secretions before and after the initiation of highly active antiretroviral therapy. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristine B Patterson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Gruber CJ, Tschugguel W, Schneeberger C, Huber JC. Production and actions of estrogens. N Engl J Med. 2002 Jan 31;346(5):340-52. doi: 10.1056/NEJMra000471. No abstract available. PMID 11821512
- [Background] Burger HG, Dudley E, Mamers P, Robertson D, Groome N, Dennerstein L. The ageing female reproductive axis I. Novartis Found Symp. 2002;242:161-7; discussion 167-71. PMID 11855686
- [Background] Gracia CR, Sammel MD, Freeman EW, Lin H, Langan E, Kapoor S, Nelson DB. Defining menopause status: creation of a new definition to identify the early changes of the menopausal transition. Menopause. 2005 Mar;12(2):128-35. doi: 10.1097/00042192-200512020-00005. PMID 15772558
- [Background] Landgren BM, Collins A, Csemiczky G, Burger HG, Baksheev L, Robertson DM. Menopause transition: Annual changes in serum hormonal patterns over the menstrual cycle in women during a nine-year period prior to menopause. J Clin Endocrinol Metab. 2004 Jun;89(6):2763-9. doi: 10.1210/jc.2003-030824. PMID 15181055
- [Background] Burger HG, Dudley EC, Robertson DM, Dennerstein L. Hormonal changes in the menopause transition. Recent Prog Horm Res. 2002;57:257-75. doi: 10.1210/rp.57.1.257. PMID 12017547
- [Background] Gracia CR, Freeman EW. Acute consequences of the menopausal transition: the rise of common menopausal symptoms. Endocrinol Metab Clin North Am. 2004 Dec;33(4):675-89. doi: 10.1016/j.ecl.2004.07.003. PMID 15501640
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] CDC HIV/AIDS Surveillance Report 2005. http://www.cdc.gov/hiv/topics/surveillance/resources/reports/index.htm#surveillance. Accessed March 8, 2007.
- [Background] Pilcher CD, Eron JJ Jr, Vemazza PL, Battegay M, Harr T, Yerly S, Vom S, Perrin L. Sexual transmission during the incubation period of primary HIV infection. JAMA. 2001 Oct 10;286(14):1713-4. doi: 10.1001/jama.286.14.1713. No abstract available. PMID 11594895
- [Background] Pedraza MA, del Romero J, Roldan F, Garcia S, Ayerbe MC, Noriega AR, Alcami J. Heterosexual transmission of HIV-1 is associated with high plasma viral load levels and a positive viral isolation in the infected partner. J Acquir Immune Defic Syndr. 1999 Jun 1;21(2):120-5. PMID 10360803
- [Background] Ragni MV, Faruki H, Kingsley LA. Heterosexual HIV-1 transmission and viral load in hemophilic patients. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Jan 1;17(1):42-5. doi: 10.1097/00042560-199801010-00006. PMID 9436757
- [Background] Quinn TC, Wawer MJ, Sewankambo N, Serwadda D, Li C, Wabwire-Mangen F, Meehan MO, Lutalo T, Gray RH. Viral load and heterosexual transmission of human immunodeficiency virus type 1. Rakai Project Study Group. N Engl J Med. 2000 Mar 30;342(13):921-9. doi: 10.1056/NEJM200003303421303. PMID 10738050
- [Background] Chakraborty H, Sen PK, Helms RW, Vernazza PL, Fiscus SA, Eron JJ, Patterson BK, Coombs RW, Krieger JN, Cohen MS. Viral burden in genital secretions determines male-to-female sexual transmission of HIV-1: a probabilistic empiric model. AIDS. 2001 Mar 30;15(5):621-7. doi: 10.1097/00002030-200103300-00012. PMID 11317000
- [Background] Royce RA, Sena A, Cates W Jr, Cohen MS. Sexual transmission of HIV. N Engl J Med. 1997 Apr 10;336(15):1072-8. doi: 10.1056/NEJM199704103361507. No abstract available. PMID 9091805
- [Background] Mofenson LM, Lambert JS, Stiehm ER, Bethel J, Meyer WA 3rd, Whitehouse J, Moye J Jr, Reichelderfer P, Harris DR, Fowler MG, Mathieson BJ, Nemo GJ. Risk factors for perinatal transmission of human immunodeficiency virus type 1 in women treated with zidovudine. Pediatric AIDS Clinical Trials Group Study 185 Team. N Engl J Med. 1999 Aug 5;341(6):385-93. doi: 10.1056/NEJM199908053410601. PMID 10432323
- [Background] Tovanabutra S, Robison V, Wongtrakul J, Sennum S, Suriyanon V, Kingkeow D, Kawichai S, Tanan P, Duerr A, Nelson KE. Male viral load and heterosexual transmission of HIV-1 subtype E in northern Thailand. J Acquir Immune Defic Syndr. 2002 Mar 1;29(3):275-83. doi: 10.1097/00126334-200203010-00008. PMID 11873077
- [Background] Fideli US, Allen SA, Musonda R, Trask S, Hahn BH, Weiss H, Mulenga J, Kasolo F, Vermund SH, Aldrovandi GM. Virologic and immunologic determinants of heterosexual transmission of human immunodeficiency virus type 1 in Africa. AIDS Res Hum Retroviruses. 2001 Jul 1;17(10):901-10. doi: 10.1089/088922201750290023. PMID 11461676
- [Background] Coombs RW, Reichelderfer PS, Landay AL. Recent observations on HIV type-1 infection in the genital tract of men and women. AIDS. 2003 Mar 7;17(4):455-80. doi: 10.1097/00002030-200303070-00001. No abstract available. PMID 12598766
- [Background] Pereira AS, Kashuba AD, Fiscus SA, Hall JE, Tidwell RR, Troiani L, Dunn JA, Eron JJ Jr, Cohen MS. Nucleoside analogues achieve high concentrations in seminal plasma: relationship between drug concentration and virus burden. J Infect Dis. 1999 Dec;180(6):2039-43. doi: 10.1086/315149. PMID 10558966
- [Background] Vernazza PL, Troiani L, Flepp MJ, Cone RW, Schock J, Roth F, Boggian K, Cohen MS, Fiscus SA, Eron JJ. Potent antiretroviral treatment of HIV-infection results in suppression of the seminal shedding of HIV. The Swiss HIV Cohort Study. AIDS. 2000 Jan 28;14(2):117-21. doi: 10.1097/00002030-200001280-00006. PMID 10708281
- [Background] Kotler DP, Shimada T, Snow G, Winson G, Chen W, Zhao M, Inada Y, Clayton F. Effect of combination antiretroviral therapy upon rectal mucosal HIV RNA burden and mononuclear cell apoptosis. AIDS. 1998 Apr 16;12(6):597-604. doi: 10.1097/00002030-199806000-00008. PMID 9583599
- [Background] Al-Harthi L, Kovacs A, Coombs RW, Reichelderfer PS, Wright DJ, Cohen MH, Cohn J, Cu-Uvin S, Watts H, Lewis S, Beckner S, Landay A; WHS 001 Study Team. A menstrual cycle pattern for cytokine levels exists in HIV-positive women: implication for HIV vaginal and plasma shedding. AIDS. 2001 Aug 17;15(12):1535-43. doi: 10.1097/00002030-200108170-00011. PMID 11504986
- [Background] Cummins JE, Christensen L, Lennox JL, Bush TJ, Wu Z, Malamud D, Evans-Strickfaden T, Siddig A, Caliendo AM, Hart CE, Dezzutti CS. Mucosal innate immune factors in the female genital tract are associated with vaginal HIV-1 shedding independent of plasma viral load. AIDS Res Hum Retroviruses. 2006 Aug;22(8):788-95. doi: 10.1089/aid.2006.22.788. PMID 16910835
- [Background] Bebell L, Passmore J, Williamson C, et al. Clincial correlations of inflammatory cytokines in the female genital tract during acute HIV-1 infection. Paper presented at: 16th International AIDS Conference, 2006; Toronto, Canada.
- [Background] Reichelderfer PS, Coombs RW, Wright DJ, Cohn J, Burns DN, Cu-Uvin S, Baron PA, Coheng MH, Landay AL, Beckner SK, Lewis SR, Kovacs AA. Effect of menstrual cycle on HIV-1 levels in the peripheral blood and genital tract. WHS 001 Study Team. AIDS. 2000 Sep 29;14(14):2101-7. doi: 10.1097/00002030-200009290-00005. PMID 11061650
- [Background] Nelson KE, Celentano DD, Suprasert S, Wright N, Eiumtrakul S, Tulvatana S, Matanasarawoot A, Akarasewi P, Kuntolbutra S, Romyen S, et al. Risk factors for HIV infection among young adult men in northern Thailand. JAMA. 1993 Aug 25;270(8):955-60. PMID 8345647
- [Background] Nicolosi A, Correa Leite ML, Musicco M, Arici C, Gavazzeni G, Lazzarin A. The efficiency of male-to-female and female-to-male sexual transmission of the human immunodeficiency virus: a study of 730 stable couples. Italian Study Group on HIV Heterosexual Transmission. Epidemiology. 1994 Nov;5(6):570-5. doi: 10.1097/00001648-199411000-00003. PMID 7841237
- [Background] Mastro TD, Satten GA, Nopkesorn T, Sangkharomya S, Longini IM Jr. Probability of female-to-male transmission of HIV-1 in Thailand. Lancet. 1994 Jan 22;343(8891):204-7. doi: 10.1016/s0140-6736(94)90990-3. PMID 7904668
- [Background] Nagot N, Ouedraogo A, Foulongne V, Konate I, Weiss HA, Vergne L, Defer MC, Djagbare D, Sanon A, Andonaba JB, Becquart P, Segondy M, Vallo R, Sawadogo A, Van de Perre P, Mayaud P; ANRS 1285 Study Group. Reduction of HIV-1 RNA levels with therapy to suppress herpes simplex virus. N Engl J Med. 2007 Feb 22;356(8):790-9. doi: 10.1056/NEJMoa062607. PMID 17314338
- [Background] Ouedraogo A, Nagot N, Vergne L, Konate I, Weiss HA, Defer MC, Foulongne V, Sanon A, Andonaba JB, Segondy M, Mayaud P, Van de Perre P. Impact of suppressive herpes therapy on genital HIV-1 RNA among women taking antiretroviral therapy: a randomized controlled trial. AIDS. 2006 Nov 28;20(18):2305-13. doi: 10.1097/QAD.0b013e328010238d. PMID 17117016
- [Background] Nagot N, Foulongne V, Becquart P, Mayaud P, Konate I, Ouedraogo A, Defer MC, Weiss H, Van de Perre P, Segondy M. Longitudinal assessment of HIV-1 and HSV-2 shedding in the genital tract of West African women. J Acquir Immune Defic Syndr. 2005 Aug 15;39(5):632-4. PMID 16044019
- [Background] Mcclelland RS, Wang CC, Mandaliya K, Overbaugh J, Reiner MT, Panteleeff DD, Lavreys L, Ndinya-Achola J, Bwayo JJ, Kreiss JK. Treatment of cervicitis is associated with decreased cervical shedding of HIV-1. AIDS. 2001 Jan 5;15(1):105-10. doi: 10.1097/00002030-200101050-00015. PMID 11192850
- [Background] St John E, Mares D, Spear GT. Bacterial vaginosis and host immunity. Curr HIV/AIDS Rep. 2007 Feb;4(1):22-8. doi: 10.1007/s11904-007-0004-y. PMID 17338857
- [Background] Sha BE, Zariffard MR, Wang QJ, Chen HY, Bremer J, Cohen MH, Spear GT. Female genital-tract HIV load correlates inversely with Lactobacillus species but positively with bacterial vaginosis and Mycoplasma hominis. J Infect Dis. 2005 Jan 1;191(1):25-32. doi: 10.1086/426394. Epub 2004 Dec 2. PMID 15592999
- [Background] Bukusi EA, Cohen CR, Meier AS, Waiyaki PG, Nguti R, Njeri JN, Holmes KK. Bacterial vaginosis: risk factors among Kenyan women and their male partners. Sex Transm Dis. 2006 Jun;33(6):361-7. doi: 10.1097/01.olq.0000200551.07573.df. PMID 16547451
- [Background] Branson BM, Handsfield HH, Lampe MA, Janssen RS, Taylor AW, Lyss SB, Clark JE; Centers for Disease Control and Prevention (CDC). Revised recommendations for HIV testing of adults, adolescents, and pregnant women in health-care settings. MMWR Recomm Rep. 2006 Sep 22;55(RR-14):1-17; quiz CE1-4. PMID 16988643
- [Background] Matthias RE, Lubben JE, Atchison KA, Schweitzer SO. Sexual activity and satisfaction among very old adults: results from a community-dwelling Medicare population survey. Gerontologist. 1997 Feb;37(1):6-14. doi: 10.1093/geront/37.1.6. PMID 9046699
- [Background] Patel D, Gillespie B, Foxman B. Sexual behavior of older women: results of a random-digit-dialing survey of 2,000 women in the United States. Sex Transm Dis. 2003 Mar;30(3):216-20. doi: 10.1097/00007435-200303000-00008. PMID 12616139
- [Background] Gott CM. Sexual activity and risk-taking in later life. Health Soc Care Community. 2001 Mar;9(2):72-8. doi: 10.1046/j.1365-2524.2001.00285.x. PMID 11560723
- [Background] Gleiter CH, Gundert-Remy U. Gender differences in pharmacokinetics. Eur J Drug Metab Pharmacokinet. 1996 Apr-Jun;21(2):123-8. doi: 10.1007/BF03190260. PMID 8839685
- [Background] Vahl N, Moller N, Lauritzen T, Christiansen JS, Jorgensen JO. Metabolic effects and pharmacokinetics of a growth hormone pulse in healthy adults: relation to age, sex, and body composition. J Clin Endocrinol Metab. 1997 Nov;82(11):3612-8. doi: 10.1210/jcem.82.11.4388. PMID 9360515
- [Background] Kishino S, Nomura A, Itoh S, Nakagawa T, Takekuma Y, Sugawara M, Furukawa H, Todo S, Miyazaki K. Age- and gender-related differences in carbohydrate concentrations of alpha1-acid glycoprotein variants and the effects of glycoforms on their drug-binding capacities. Eur J Clin Pharmacol. 2002 Dec;58(9):621-8. doi: 10.1007/s00228-002-0530-x. Epub 2002 Nov 22. PMID 12483455
- [Background] Tuck CH, Holleran S, Berglund L. Hormonal regulation of lipoprotein(a) levels: effects of estrogen replacement therapy on lipoprotein(a) and acute phase reactants in postmenopausal women. Arterioscler Thromb Vasc Biol. 1997 Sep;17(9):1822-9. doi: 10.1161/01.atv.17.9.1822. PMID 9327783
- [Background] Columbo S, Buclin T, Decosterd L, al. e. Orosmucoid plasma concentrations and genetic variants: effects on protease inhibitor clearance and cellular accumulation ratio. Paper presented at: 7th International Workshop on Clinical Pharmacology of HIV Therapy; April 20-22, 2006, 2006; Lisbon, Portugal.
- [Background] Barry M, Gibbons S, Back D, Mulcahy F. Protease inhibitors in patients with HIV disease. Clinically important pharmacokinetic considerations. Clin Pharmacokinet. 1997 Mar;32(3):194-209. doi: 10.2165/00003088-199732030-00003. PMID 9084959
- [Background] Hashimoto S, Miwa M, Akasofu K, Nishida E. Changes in 40 serum proteins of post-menopausal women. Maturitas. 1991 Mar;13(1):23-33. doi: 10.1016/0378-5122(91)90282-u. PMID 1861640
- [Background] Baker SD, Grochow LB. Pharmacology of cancer chemotherapy in the older person. Clin Geriatr Med. 1997 Feb;13(1):169-83. PMID 8995106
- [Background] Egorin MJ. Cancer pharmacology in the elderly. Semin Oncol. 1993 Feb;20(1):43-9. No abstract available. PMID 8475409
- [Background] Grandison MK, Boudinot FD. Age-related changes in protein binding of drugs: implications for therapy. Clin Pharmacokinet. 2000 Mar;38(3):271-90. doi: 10.2165/00003088-200038030-00005. PMID 10749520
- [Background] Krecic-Shepard ME, Barnas CR, Slimko J, Schwartz JB. Faster clearance of sustained release verapamil in men versus women: continuing observations on sex-specific differences after oral administration of verapamil. Clin Pharmacol Ther. 2000 Sep;68(3):286-92. doi: 10.1067/mcp.2000.109356. PMID 11014410
- [Background] Schuetz EG, Furuya KN, Schuetz JD. Interindividual variation in expression of P-glycoprotein in normal human liver and secondary hepatic neoplasms. J Pharmacol Exp Ther. 1995 Nov;275(2):1011-8. PMID 7473127
- [Background] Krecic-Shepard ME, Barnas CR, Slimko J, Jones MP, Schwartz JB. Gender-specific effects on verapamil pharmacokinetics and pharmacodynamics in humans. J Clin Pharmacol. 2000 Mar;40(3):219-30. doi: 10.1177/00912700022008883. PMID 10709150
- [Background] Krecic-Shepard ME, Park K, Barnas C, Slimko J, Kerwin DR, Schwartz JB. Race and sex influence clearance of nifedipine: results of a population study. Clin Pharmacol Ther. 2000 Aug;68(2):130-42. doi: 10.1067/mcp.2000.108678. PMID 10976544
- [Background] Kharasch ED, Mautz D, Senn T, Lentz G, Cox K. Menstrual cycle variability in midazolam pharmacokinetics. J Clin Pharmacol. 1999 Mar;39(3):275-80. PMID 10073327
- [Background] Kosel BW, Beckerman KP, Hayashi S, Homma M, Aweeka FT. Pharmacokinetics of nelfinavir and indinavir in HIV-1-infected pregnant women. AIDS. 2003 May 23;17(8):1195-9. doi: 10.1097/00002030-200305230-00011. PMID 12819521
- [Background] Acosta EP, Zorrilla C, Van Dyke R, Bardeguez A, Smith E, Hughes M, Huang S, Pitt J, Watts H, Mofenson L; Pediatric AIDS Clinical Trials Group 386 Protocol Team. Pharmacokinetics of saquinavir-SGC in HIV-infected pregnant women. HIV Clin Trials. 2001 Nov-Dec;2(6):460-5. doi: 10.1310/PUY3-5JWL-FX2B-98VU. PMID 11742433
- [Background] Abernethy DR, Greenblatt DJ, Shader RI. Imipramine and desipramine disposition in the elderly. J Pharmacol Exp Ther. 1985 Jan;232(1):183-8. PMID 3965690
- [Background] Dahl ML, Bertilsson L, Nordin C. Steady-state plasma levels of nortriptyline and its 10-hydroxy metabolite: relationship to the CYP2D6 genotype. Psychopharmacology (Berl). 1996 Feb;123(4):315-9. doi: 10.1007/BF02246640. PMID 8867869
- [Background] Walle UK, Fagan TC, Topmiller MJ, Conradi EC, Walle T. The influence of gender and sex steroid hormones on the plasma binding of propranolol enantiomers. Br J Clin Pharmacol. 1994 Jan;37(1):21-5. doi: 10.1111/j.1365-2125.1994.tb04233.x. PMID 8148214
- [Background] Wadelius M, Darj E, Frenne G, Rane A. Induction of CYP2D6 in pregnancy. Clin Pharmacol Ther. 1997 Oct;62(4):400-7. doi: 10.1016/S0009-9236(97)90118-1. PMID 9357391
- [Background] Aldridge A, Bailey J, Neims AH. The disposition of caffeine during and after pregnancy. Semin Perinatol. 1981 Oct;5(4):310-4. No abstract available. PMID 7302604
- [Background] Knutti R, Rothweiler H, Schlatter C. Effect of pregnancy on the pharmacokinetics of caffeine. Eur J Clin Pharmacol. 1981;21(2):121-6. doi: 10.1007/BF00637512. PMID 7341280
- [Background] Kalow W, Tang BK. Use of caffeine metabolite ratios to explore CYP1A2 and xanthine oxidase activities. Clin Pharmacol Ther. 1991 Nov;50(5 Pt 1):508-19. doi: 10.1038/clpt.1991.176. PMID 1934864
- [Background] Ou-Yang DS, Huang SL, Wang W, Xie HG, Xu ZH, Shu Y, Zhou HH. Phenotypic polymorphism and gender-related differences of CYP1A2 activity in a Chinese population. Br J Clin Pharmacol. 2000 Feb;49(2):145-51. doi: 10.1046/j.1365-2125.2000.00128.x. PMID 10671909
- [Background] Relling MV, Lin JS, Ayers GD, Evans WE. Racial and gender differences in N-acetyltransferase, xanthine oxidase, and CYP1A2 activities. Clin Pharmacol Ther. 1992 Dec;52(6):643-58. doi: 10.1038/clpt.1992.203. PMID 1458773
- [Background] Tamminga WJ, Wemer J, Oosterhuis B, Weiling J, Wilffert B, de Leij LF, de Zeeuw RA, Jonkman JH. CYP2D6 and CYP2C19 activity in a large population of Dutch healthy volunteers: indications for oral contraceptive-related gender differences. Eur J Clin Pharmacol. 1999 May;55(3):177-84. doi: 10.1007/s002280050615. PMID 10379632
- [Background] Tamminga WJ, Wemer J, Oosterhuis B, de Zeeuw RA, de Leij LF, Jonkman JH. The prevalence of CYP2D6 and CYP2C19 genotypes in a population of healthy Dutch volunteers. Eur J Clin Pharmacol. 2001 Dec;57(10):717-22. doi: 10.1007/s002280100359. PMID 11829201
- [Background] Laine K, Tybring G, Bertilsson L. No sex-related differences but significant inhibition by oral contraceptives of CYP2C19 activity as measured by the probe drugs mephenytoin and omeprazole in healthy Swedish white subjects. Clin Pharmacol Ther. 2000 Aug;68(2):151-9. doi: 10.1067/mcp.2000.108949. PMID 10976546
- [Background] Toornvliet R, van Berckel BN, Luurtsema G, Lubberink M, Geldof AA, Bosch TM, Oerlemans R, Lammertsma AA, Franssen EJ. Effect of age on functional P-glycoprotein in the blood-brain barrier measured by use of (R)-[(11)C]verapamil and positron emission tomography. Clin Pharmacol Ther. 2006 Jun;79(6):540-8. doi: 10.1016/j.clpt.2006.02.004. PMID 16765142
- [Background] Fleishaker JC, Pearson LK, Pearson PG, Wienkers LC, Hopkins NK, Peters GR. Hormonal effects on tirilazad clearance in women: assessment of the role of CYP3A. J Clin Pharmacol. 1999 Mar;39(3):260-7. PMID 10073325
- [Background] Harris RZ, Tsunoda SM, Mroczkowski P, Wong H, Benet LZ. The effects of menopause and hormone replacement therapies on prednisolone and erythromycin pharmacokinetics. Clin Pharmacol Ther. 1996 Apr;59(4):429-35. doi: 10.1016/S0009-9236(96)90112-5. PMID 8612388
- [Background] Lemmens HJ, Burm AG, Hennis PJ, Gladines MP, Bovill JG. Influence of age on the pharmacokinetics of alfentanil. Gender dependence. Clin Pharmacokinet. 1990 Nov;19(5):416-22. doi: 10.2165/00003088-199019050-00005. PMID 2268988
- [Background] Rubio A, Cox C. Sex, age and alfentanil pharmacokinetics. Clin Pharmacokinet. 1991 Jul;21(1):81-2. doi: 10.2165/00003088-199121010-00006. No abstract available. PMID 1914343
- [Background] Muck W. Clinical pharmacokinetics of cerivastatin. Clin Pharmacokinet. 2000 Aug;39(2):99-116. doi: 10.2165/00003088-200039020-00002. PMID 10976657
- [Background] Miners JO, Robson RA, Birkett DJ. Gender and oral contraceptive steroids as determinants of drug glucuronidation: effects on clofibric acid elimination. Br J Clin Pharmacol. 1984 Aug;18(2):240-3. doi: 10.1111/j.1365-2125.1984.tb02461.x. PMID 6487463
- [Background] Kashuba AD, Bertino JS Jr, Kearns GL, Leeder JS, James AW, Gotschall R, Nafziger AN. Quantitation of three-month intraindividual variability and influence of sex and menstrual cycle phase on CYP1A2, N-acetyltransferase-2, and xanthine oxidase activity determined with caffeine phenotyping. Clin Pharmacol Ther. 1998 May;63(5):540-51. doi: 10.1016/S0009-9236(98)90105-9. PMID 9630827
- [Background] Macdonald JI, Herman RJ, Verbeeck RK. Sex-difference and the effects of smoking and oral contraceptive steroids on the kinetics of diflunisal. Eur J Clin Pharmacol. 1990;38(2):175-9. doi: 10.1007/BF00265980. PMID 2338115
- [Background] Brenner BM, Meyer TW, Hostetter TH. Dietary protein intake and the progressive nature of kidney disease: the role of hemodynamically mediated glomerular injury in the pathogenesis of progressive glomerular sclerosis in aging, renal ablation, and intrinsic renal disease. N Engl J Med. 1982 Sep 9;307(11):652-9. doi: 10.1056/NEJM198209093071104. No abstract available. PMID 7050706
- [Background] James GD, Sealey JE, Alderman M, Ljungman S, Mueller FB, Pecker MS, Laragh JH. A longitudinal study of urinary creatinine and creatinine clearance in normal subjects. Race, sex, and age differences. Am J Hypertens. 1988 Apr;1(2):124-31. doi: 10.1093/ajh/1.2.124. PMID 3401350
- [Background] Anderson PL, Kakuda TN, Kawle S, Fletcher CV. Antiviral dynamics and sex differences of zidovudine and lamivudine triphosphate concentrations in HIV-infected individuals. AIDS. 2003 Oct 17;17(15):2159-68. doi: 10.1097/00002030-200310170-00003. PMID 14523272
- [Background] Stretcher BN, Pesce AJ, Frame PT, Stein DS. Pharmacokinetics of zidovudine phosphorylation in peripheral blood mononuclear cells from patients infected with human immunodeficiency virus. Antimicrob Agents Chemother. 1994 Jul;38(7):1541-7. doi: 10.1128/AAC.38.7.1541. PMID 7979286
- [Background] Harris M, Back D, Kewn S, Jutha S, Marina R, Montaner JS. Intracellular carbovir triphosphate levels in patients taking abacavir once a day. AIDS. 2002 May 24;16(8):1196-7. doi: 10.1097/00002030-200205240-00021. No abstract available. PMID 12004286
- [Background] Green D, Jonusas A, Montague JR, Mudd LM. Tyrosine kinase activity of nerve growth factor and estrogen in embryonic septal neurons cultured from the rat. Neurochem Res. 2002 Dec;27(12):1699-705. doi: 10.1023/a:1021651530846. PMID 12515325
- [Background] Cui Y, Parra I, Zhang M, Hilsenbeck SG, Tsimelzon A, Furukawa T, Horii A, Zhang ZY, Nicholson RI, Fuqua SA. Elevated expression of mitogen-activated protein kinase phosphatase 3 in breast tumors: a mechanism of tamoxifen resistance. Cancer Res. 2006 Jun 1;66(11):5950-9. doi: 10.1158/0008-5472.CAN-05-3243. PMID 16740736
- [Background] Muraki K, Okuya S, Tanizawa Y. Estrogen receptor alpha regulates insulin sensitivity through IRS-1 tyrosine phosphorylation in mature 3T3-L1 adipocytes. Endocr J. 2006 Dec;53(6):841-51. doi: 10.1507/endocrj.k06-005. Epub 2006 Sep 26. PMID 17001108
- [Background] Burger D, van der Heiden I, la Porte C, van der Ende M, Groeneveld P, Richter C, Koopmans P, Kroon F, Sprenger H, Lindemans J, Schenk P, van Schaik R. Interpatient variability in the pharmacokinetics of the HIV non-nucleoside reverse transcriptase inhibitor efavirenz: the effect of gender, race, and CYP2B6 polymorphism. Br J Clin Pharmacol. 2006 Feb;61(2):148-54. doi: 10.1111/j.1365-2125.2005.02536.x. PMID 16433869
- [Background] Gatti G, dePascalis C, deLucca A. Predictors of amprenavir parameters of drug exposure in heavily pretreated HIV positive patients. Paper presented at: Proceedings on the 6th International Congress on Drug therapy in HIV infection, 2002; Glasgow, Scotland.
- [Background] Pai MP, Schriever CA, Diaz-Linares M, Novak RM, Rodvold KA. Sex-related differences in the pharmacokinetics of once-daily saquinavir soft-gelatin capsules boosted with low-dose ritonavir in patients infected with human immunodeficiency virus type 1. Pharmacotherapy. 2004 May;24(5):592-9. doi: 10.1592/phco.24.6.592.34744. PMID 15162893
- [Background] Umeh O, Currier J, Park J, et al. Sex differences in lopinavir/ritonavir soft gel capsule pharmacokinetics among HIV-infected females and males. Paper presented at: 14th Conference on Retroviruses and Opportunistic Infections, 2007; Los Angelos, CA.
- [Background] Fletcher CV, Jiang H, Brundage RC, Acosta EP, Haubrich R, Katzenstein D, Gulick RM. Sex-based differences in saquinavir pharmacology and virologic response in AIDS Clinical Trials Group Study 359. J Infect Dis. 2004 Apr 1;189(7):1176-84. doi: 10.1086/382754. Epub 2004 Mar 16. PMID 15031785
- [Background] Burger DM, Siebers MC, Hugen PW, Aarnoutse RE, Hekster YA, Koopmans PP. Pharmacokinetic variability caused by gender: do women have higher indinavir exposure than men? J Acquir Immune Defic Syndr. 2002 Jan 1;29(1):101-2. doi: 10.1097/00126334-200201010-00014. No abstract available. PMID 11782597
- [Background] Burger D, Boyd M, Duncombe C, Felderhof M, Mahanontharit A, Ruxrungtham K, Ubolyam S, Stek M, Cooper D, Lange J, Phanupak P, Reiss P. Pharmacokinetics and pharmacodynamics of indinavir with or without low-dose ritonavir in HIV-infected Thai patients. J Antimicrob Chemother. 2003 May;51(5):1231-8. doi: 10.1093/jac/dkg198. Epub 2003 Mar 28. PMID 12668574
- [Background] Vernazza PL, Eron JJ, Fiscus SA, Cohen MS. Sexual transmission of HIV: infectiousness and prevention. AIDS. 1999 Feb 4;13(2):155-66. doi: 10.1097/00002030-199902040-00003. No abstract available. PMID 10202821
- [Background] Vernazza PL, Gilliam BL, Flepp M, Dyer JR, Frank AC, Fiscus SA, Cohen MS, Eron JJ. Effect of antiviral treatment on the shedding of HIV-1 in semen. AIDS. 1997 Aug;11(10):1249-54. doi: 10.1097/00002030-199710000-00008. PMID 9256943
- [Background] Vernazza PL, Kashuba AD, Cohen MS. Biological Correlates of Sexual Transmission of HIV Practical Consequences and Potential Targets for Public Health : Practical Consequences and Potential Targets for Public Health. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2002 Mar;45(3):277-85. doi: 10.1007/s00103-001-0367-y. PMID 24676923
- [Background] Dumond J, Yeh R, Patterson K, et al. First Dose and Steady-state Genital Tract Pharmacokinetics of Ten Antiretroviral Drugs in HIV-infected Women: Implications for Pre- and Post- Exposure Prophylaxis. Paper presented at: 13th Conference on Retroviruses and Opportunistic Infections, 2006; Denver, CO.
- [Background] Min SS, Corbett AH, Rezk N, Cu-Uvin S, Fiscus SA, Petch L, Cohen MS, Kashuba AD. Protease inhibitor and nonnucleoside reverse transcriptase inhibitor concentrations in the genital tract of HIV-1-infected women. J Acquir Immune Defic Syndr. 2004 Dec 15;37(5):1577-80. doi: 10.1097/00126334-200412150-00008. PMID 15577412
- [Background] Cohen MS, Gay C, Kashuba AD, Blower S, Paxton L. Narrative review: antiretroviral therapy to prevent the sexual transmission of HIV-1. Ann Intern Med. 2007 Apr 17;146(8):591-601. doi: 10.7326/0003-4819-146-8-200704170-00010. PMID 17438318
- [Background] Napravnik S, Poole C, Thomas JC, Eron JJ Jr. Gender difference in HIV RNA levels: a meta-analysis of published studies. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):11-9. doi: 10.1097/00126334-200209010-00002. PMID 12352145
- [Background] Fletcher CV, Acosta EP, Henry K, Page LM, Gross CR, Kawle SP, Remmel RP, Erice A, Balfour HH Jr. Concentration-controlled zidovudine therapy. Clin Pharmacol Ther. 1998 Sep;64(3):331-8. doi: 10.1016/S0009-9236(98)90182-5. PMID 9757157
- [Background] Fletcher CV, Anderson PL, Kakuda TN, Schacker TW, Henry K, Gross CR, Brundage RC. Concentration-controlled compared with conventional antiretroviral therapy for HIV infection. AIDS. 2002 Mar 8;16(4):551-60. doi: 10.1097/00002030-200203080-00006. PMID 11872998
- [Background] Reddy S, Troiani L, Pereira A, et al. Zidovudine and Lamivudine (ZDV/3TC) Seminal Plasma:Blood Plasma (SP:BP) Concentration (CONC) Ratios Do Not Predict Total SP Exposure. Paper presented at: World AIDS Conference, 2002; Barcelona, Sapin.
- [Background] Council. USDoHaHSDPoAGfAaA--AWGotOoARA. Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents. www.aidsinfo.nih.gov. Accessed March 26, 2007.
- [Background] Jung BH, Rezk NL, Bridges AS, Corbett AH, Kashuba AD. Simultaneous determination of 17 antiretroviral drugs in human plasma for quantitative analysis with liquid chromatography-tandem mass spectrometry. Biomed Chromatogr. 2007 Oct;21(10):1095-104. doi: 10.1002/bmc.865. PMID 17582235
- [Background] King T, Bushman L, Kiser J, Anderson PL, Ray M, Delahunty T, Fletcher CV. Liquid chromatography-tandem mass spectrometric determination of tenofovir-diphosphate in human peripheral blood mononuclear cells. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Nov 7;843(2):147-56. doi: 10.1016/j.jchromb.2006.05.043. Epub 2006 Jul 7. PMID 16828350
- [Background] Robbins BL, Poston PA, Neal EF, Slaughter C, Rodman JH. Simultaneous measurement of intracellular triphosphate metabolites of zidovudine, lamivudine and abacavir (carbovir) in human peripheral blood mononuclear cells by combined anion exchange solid phase extraction and LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2007 May 1;850(1-2):310-7. doi: 10.1016/j.jchromb.2006.12.015. Epub 2006 Dec 17. PMID 17197254
- [Background] Darque A, Valette G, Rousseau F, Wang LH, Sommadossi JP, Zhou XJ. Quantitation of intracellular triphosphate of emtricitabine in peripheral blood mononuclear cells from human immunodeficiency virus-infected patients. Antimicrob Agents Chemother. 1999 Sep;43(9):2245-50. doi: 10.1128/AAC.43.9.2245. PMID 10471573
- [Background] Stek AM, Mirochnick M, Capparelli E, Best BM, Hu C, Burchett SK, Elgie C, Holland DT, Smith E, Tuomala R, Cotter A, Read JS. Reduced lopinavir exposure during pregnancy. AIDS. 2006 Oct 3;20(15):1931-9. doi: 10.1097/01.aids.0000247114.43714.90. PMID 16988514
- [Background] Sadiq ST, Taylor S, Kaye S, Bennett J, Johnstone R, Byrne P, Copas AJ, Drake SM, Pillay D, Weller I. The effects of antiretroviral therapy on HIV-1 RNA loads in seminal plasma in HIV-positive patients with and without urethritis. AIDS. 2002 Jan 25;16(2):219-25. doi: 10.1097/00002030-200201250-00011. PMID 11807306